CLINICAL TRIAL: NCT06351527
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ICP-248 as Monotherapy or in Combination With Anti-CD20 Monoclonal Antibody in Patients With Mature B-cell Malignancies
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ICP-248 as Monotherapy or in Combination With Anti-CD20 Monoclonal Antibody in Mature B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InnoCare Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-01202
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Mature B-cell Malignancies
MeSH Terms: interventions — obinutuzumab; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-Escalation Cohort - CLL/SLL and MCL (Experimental): Participants will receive ICP-248 daily from an initial dose of 5/10 mg to the target dose. Cycles will comprise 28 days.
  Interventions: Drug: ICP-248
- Dose-Expansion Cohort A - CLL/SLL (Experimental): Participants will receive ICP-248 daily from an initial dose of 5/10 mg to the target dose and obinutuzumab for 6 cycles. Cycles will comprise 28 days.
  Interventions: Drug: ICP-248; Drug: Obinutuzumab (G)
- Dose-Expansion Cohort B - MCL (Experimental): Participants will receive ICP-248 daily from an initial dose of 5/10 mg to the target dose. Cycles will comprise 28 days.
  Interventions: Drug: ICP-248
- Dose-Expansion Cohort C - MCL (Experimental): Participants will receive ICP-248 daily from an initial dose of 5/10 mg to the target dose and Rituximab for 18 cycles. Cycles will comprise 28 days.
  Interventions: Drug: ICP-248; Drug: Rituximab (R)

INTERVENTIONS:
Drug: ICP-248 — ICP-248 will be administered orally once daily at escalated doses (starting dose 5/10 mg, maximum 150 mg).
Drug: Obinutuzumab (G) — Obinutuzumab will be administered by IV infusion at a dose of 100 mg or 1000 mg, depending on splitting rules, at Cycle 1, Day 1 (if 100 mg was received on Day 1, 900 mg will be administered on Cycle 1, Day 2); 1000 mg at Cycle 1, Day 8 and Day 15; 1000 mg at Day 1 for all subsequent cycles until the end of Cycle 6.
  Arms: Dose-Expansion Cohort A - CLL/SLL
Drug: Rituximab (R) — Rituximab will be administered by IV infusion at a dose of 375 milligrams per square meter (mg/m^2) at Day 1 per week for 4 weeks during cycle 1, then on day 1 of cycles 3-8, and thereafter once every other cycle up to 2 years.
  Arms: Dose-Expansion Cohort C - MCL

SUMMARY:
Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of ICP-248 as monotherapy or in combination with anti-CD20 monoclonal antibody in Mature B-cell Malignancies

ELIGIBILITY:
1. Age ≥ 18.
2. Subjects with histopathologically and/or flow cytometry-confirmed diseases according to the 2016 World Health Organization (WHO) classification criteria for lymphohematopoietic neoplasms or meeting the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria: relapsed or refractory CLL/SLL, relapsed or refractory MCL. Patients must have received at least two prior lines of adequate systemic therapy before study entry, and at least one prior systemic therapy should include Bruton's kinase inhibitor (BTKi).
3. For subjects with R/R MCL: Patients must have measurable disease per the Lugano 2014 criteria.
4. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of ≤ 1 and a life expectancy of ≥ 6 months.
5. Adequate hematologic, hepatic, renal, pulmonary and cardiac function
6. Patients with basically normal coagulation function
7. Patients with fertility potential and their partners need contraception
8. Subjects can communicate with the investigator well and to complete the study as specified in the study.

Exclusion Criteria:

1. Known central nervous system involvement by lymphoma/leukemia.
2. Known or suspected history of Richter's transformation.
3. Prior autologous stem cell transplant (unless ≥ 3 months since transplant); or prior chimeric cell therapy (unless ≥ 3 months since cell infusion).
4. A history of allogeneic stem cell transplantation.
5. An interval of less than 5 half-lives from the last dose of a strong CYP3A or CYP2C8 inhibitor or inducer (chemical agent, herbal medicine and dietary supplement) to the first dose of the investigational product, or a plan to use concurrently medications, dietary supplements or food (e.g., grapefruit or grapefruit juice) with strong CYP3A or CYP2C8 inhibitory or inductive effect during study participation
6. Presence of active infection that currently requires intravenous systemic anti-infective therapy.
7. History of immunodeficiency, including a positive human immunodeficiency virus (HIV) antibody test.
8. History of significant cardiovascular disease
9. Patients with previous or concomitant central nervous system disorders
10. Grade 2 or above toxicity due to prior anti-cancer therapy at screening
11. Known alcohol or drug dependence
12. Unable to swallow tablets or presence of disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2027-06-25 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
DLT | 49 days
  Dose-limiting toxicity (DLT) rate at each dose level DLT will be assessed via CTCAE version 5.0 or iwCLL 2018.
Safety and tolerability of ICP-248 at different doses in B-cell malignancies | 5 years
  To investigate the incidence, nature and severity of adverse events (AE) according to NCI-CTCAE V5.0 evaluation criteria or iwCLL 2018.

SECONDARY OUTCOMES:
Cmax, ss of ICP-248 | Predose up to week 28
  Steady State Maximum Concentration of ICP-248
Ctrough, ss of ICP-248 | Predose up to week 28
  Steady State Trough Concentration of ICP-248
Preliminary efficacy of ICP-248 monotherapy in patients with B-cell malignancy | 5 years
  Investigator-assessed ORR and CRR as defined by the Lugano 2014 Classification or per iwCLL 2018 criteria

CONTACTS AND LOCATIONS:
Locations (8):
- United States (2):
  - BRCR Medical Center, Plantation, Florida
  - Clinical Research Alliance, Westbury, New York
- Pan American Center for Oncology Trials, San Juan, Puerto Rico
- Ukraine (5):
  - CNE CCOHTPC of Cherkasy Regional Council, Cherkasy
  - CNE"City Clin Hosp#4"of Dnipro City Council, Dnipro
  - Medical Center of Limited Liability Company Arensia Exploratory Medicine, Kyiv
  - Med Center 'Ok!Clinic+' of International Institute of Clinical Trials LLC, Kyiv
  - SI Institute of Blood Pathology and Transfusion Medicine of AMSU, Lviv